CLINICAL TRIAL: NCT02690896
Title: Caregiver Burden and Depression: Caring for Those Who Care for Others
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: Alzheimer's and Dementia Resource Center (Unknown)
Responsible Party: Principal Investigator, Daniel Paulson, Assistant Professor, University of Central Florida
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBE-15-11548
Record Dates: First submitted 2016-01-11; First posted 2016-02-24 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Dementia; Alzheimer's Disease
Keywords: caregiver burden; caregiver support groups
MeSH Terms: conditions — Dementia; Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UCF Behavioral Intervention Group (Experimental): The intervention group will be the UCF Caregiver Support. Participants will receive a 90 minute group session, once a week, for a period of 6 consecutive weeks.
  Interventions: Behavioral: UCF Caregiver Support Group
- Community Comparison Group (Active Comparator): Comparison group members will come from potential local support groups include, but are not limited to, the support group at the Faith Assembly of God church, the caregiver support group at the First Baptist Church of Orlando, and the caregiver support group at the Alzheimer's and Dementia Resource Center.
  Interventions: Behavioral: Community Support Groups

INTERVENTIONS:
Behavioral: UCF Caregiver Support Group — The intervention will be a 90 minute group session, once a week, for a period of 6 consecutive weeks. The intervention will teach caregivers specific behavioral techniques for managing care recipients' symptoms in the home environment and encourage caregiver self-care.
  Arms: UCF Behavioral Intervention Group
Behavioral: Community Support Groups — Comparison group members will come from local community support groups, which typically include components of social support and limited psychoeducation, and are relatively unstructured.
  Arms: Community Comparison Group

SUMMARY:
The purpose of this study is to examine the effectiveness of support group intervention for primary caregivers of a person with dementia or similar cognitive impairment.

DETAILED DESCRIPTION:
This research aims to determine if participation in caregiver support groups and individual differences between caregivers influence the decision of the caregiver to place their family member in a long-term care facility. This research also aims to identify significant predictor variables of outcome. The intervention to be employed has been empirically supported by past research (Gonyea, 2006), but additional research is required to establish this intervention as an empirically supported treatment for caregivers. The proposed research will examine the hypotheses that: (A) a brief 6-session caregiver support group will reduce caregiver burden and depression and delay or prevent transition to long-term care (e.g., nursing home care); and (B) specific caregiver characteristics will emerge as significant moderators of treatment outcomes.

The first activity of the proposed research will involve the advertisement of the caregiver support group. The caregiver support group advertisement will be posted in various facilities related to the care of older adults in the surrounding community and will also be distributed via email listserves. Next, individuals who are interested in the study and caregiver support group will contact the principal investigator or research assistants via the telephone number or email address listed on the advertisement. The proposed research utilizes a UCF behavioral intervention group and a community comparison group. The UCF behavioral intervention group will be based on the principles of behavior therapy and behavioral activation. Groups are designed to teach caregivers specific behavioral techniques for managing care recipients' symptoms in the home environment. The community comparison group will be a "treatment as usual" group; participants will be recruited from various established caregiver support groups in the community. The UCF behavioral intervention caregiver support groups will be highly structured and will be conducted with up to 13 members. The UCF behavioral intervention caregiver support groups will be run over the course of 6 weeks, with groups meeting once a week for 90 minutes. Groups will be scheduled at weekly intervals, as is characteristic for most psychotherapeutic support groups. The intake packet will include questions that are biological, psychological, and social in nature. Caregivers will also be asked questions related to their caregiving situation. Included in the packet are the following measures: demographic survey, ADL and IADL survey, caregiver preparedness scale, Center for Epidemiological Studies Short Depression Scale (CES-D 10), familial obligation scale, caregiver strain index, a neuropsychological symptom index, and a satisfaction survey. In addition, participants will completed at-home collection of saliva samples for measurement of stress hormone variation (cortisol). Saliva samples will be collected using oral swabs, which will be stored in number-coded tubes. Participants will record the time of day samples were collected, and provide subjective measures of psychological stress. Completed sample kits will be collected by study research assistants and brought back to th lab freezer for storage. This procedure will be repeated after the final session of the intervention. The group facilitator and co-faclitator will review the consent form with caregivers in person at the beginning of the first session. Participants who agree to take part in the caregiver support group and the proposed research will be given a copy of the consent form and will remain present for the current and subsequent sessions. If a participant is absent from a UCF behavioral intervention group session, he/she will be contacted by telephone and encouraged to attend future session as is consistent with standard clinic procedure. The investigators will not exclude a participant's data from analyses if he/she does not attend all six sessions.

Participants will be audio taped during this study. If a participant does not want to be audio taped, he/she will not be able to participate in the study and will be referred to an alternate provider if interested in receiving services elsewhere. The purpose of audio taping is to monitor consistency among the group sessions and to ensure treatment fidelity. The recordings will be reviewed only by principle investigator Dr. Paulson and the co-investigators, and will be deleted within two weeks of the recording. Audio recordings will be saved locally on an encrypted iPad used only for research purposes that is stored in a locked file cabinet in the OLDeR research lab, which requires code and card access.

Follow-up will be performed at 6 month intervals until the caregiving relationship has ended (if the caregiving relationship persists, follow-up will cease at 5 years).

For both the UCF behavioral intervention group and the community comparison group, participants will be contacted via telephone at 6 month intervals (after the termination of the 6-week support group for the UCF behavioral intervention group, and every 6 months following the termination of the first UCF behavioral intervention caregiver support group for community comparison participants).

The intended sample size for the proposed research includes 30 participants in the UCF behavioral intervention group and 30 participants in the community comparison group for a total of 60 participants.

Proposed statistical methods for data analyses include intent-to-treat (ITT) with last observation carried forward.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be currently providing care to a demented or cognitively impaired adult
* All participants must live in the United States.
* Participants in the community comparison group must be currently enrolled in a caregiver support group in the community (i.e., not the UCF caregiver support group).

Exclusion Criteria:

- Participants who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Long-Term Care Utilization based on Caregiver Report | baseline, 6 weeks, and then every 6 months for 5 years
  Caregivers will be asked where there care recipient lives at baseline, and then their current living status thereafter to know if and when a transition to a long-term care facility occurs.

SECONDARY OUTCOMES:
Neuropsychiatric symptoms | baseline, 6 weeks, and then every 6 months for 5 years
  Caregivers will provide an assessment of their care recipient's neuropsychiatric functioning by completing the Neuropsychiatric Inventory.
Caregiver strain | baseline, 6 weeks, and then every 6 months for 5 years
  Caregivers will provide an assessment of the burden associated with caregiving that they experience by completing The Caregiver Strain Index.
Caregiver depression | baseline, 6 weeks, and then every 6 months for 5 years
  Caregiver depression will assessed by the Center for Epidemiologic Studies Short Depression Scale (CESD-10).
Caregiver preparedness | baseline, 6 weeks, and then every 6 months for 5 years
  Caregivers will complete the The Preparedness for Caregiving Scale to assess how prepared they feel to perform the various aspects of caregiving.
Satisfaction Survey | at 6 weeks
  Participants in the UCF Caregiver Support Group will also complete a group satisfaction survey during the last session (week 6) to determine how effective they felt the group intervention is.
Stress hormone level | at baseline and 6 weeks
  Stress hormone level will be measured by cortisol levels obtained via saliva samples. Saliva samples will be collected via oral swabs for two consecutive days at both the morning and evening hours, at baseline and 6 weeks.
Daily stress inventory | at baseline and 6 weeks
  Daily stress will be measured using the Daily Inventory of Stressful Events to assess subjective psychological stress experienced.
Subjective stress | at baseline and 6 weeks
  The Pre-water Stress VAS will be used as another subjective measure of psychological stress experienced.
Emotional affective state | at baseline and 6 weeks
  The Positive and Negative Affect Schedule (PANAS) will be used as another subjective measure of psychological stress experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Paulson, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonyea JG, O'Connor MK, Boyle PA. Project CARE: a randomized controlled trial of a behavioral intervention group for Alzheimer's disease caregivers. Gerontologist. 2006 Dec;46(6):827-32. doi: 10.1093/geront/46.6.827. PMID 17169938
- See also: Please contact the UCF OLDeR Lab for any questions regarding the study and/or study materials. — http://psychology.cos.ucf.edu/older/
- Available data/document: Study-related materials — http://psychology.cos.ucf.edu/older/ — Please contact the UCF OLDeR Lab for any questions regarding the study and/or study materials.